CLINICAL TRIAL: NCT06210126
Title: Effect of Pectointercostal Fascial Plane (PIF) Block on Postoperative Chronic Pain in Patients Undergoing Open Heart Surgery: Randomized, Controlled Study
Brief Title: Pectointercostal Fascial Plane Block Chronic Pain Sternotomy
Acronym: PIFB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Betul Kozanhan, Prof. Dr, Konya Meram State Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 12-31
Record Dates: First submitted 2023-12-20; First posted 2024-01-18 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Anesthetics, Local

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pectointercostal Fascial Plane Block Group (Active Comparator): In addition to routine standard perioperative and postoperative analgesia protocol patients will receive bilateral local anesthetic injections at the Pectointercostal Fascial Plane Block
  Interventions: Other: local anesthetic injection
- Control (Other): Patients will receive standard perioperative and postoperative analgesia protocol
  Interventions: Other: Standard perioperative and postoperative analgesia protocol

INTERVENTIONS:
Other: local anesthetic injection — Ultrasound-guided pectointercostal fascial plane block group using 20 mL of 0.25% bupivacaine
  Arms: Pectointercostal Fascial Plane Block Group
Other: Standard perioperative and postoperative analgesia protocol — postoperative IV morphine PCA and paracetamol will be given. If VAS is 3 or above, 75 mg dexketoprofen trometamol will be administered.
  Arms: Control

SUMMARY:
This study aims to compare the effect of pectointercostal fascial plane block (PIFB) on postoperative chronic pain in patients undergoing open heart surgery with the standard multimodal analgesia technique.

DETAILED DESCRIPTION:
Chronic postsurgical pain (CPSP), defined as persistent pain at the surgical site or referred areas lasting at least three months post-surgery, poses a considerable challenge, notably after median sternotomy in cardiac procedures. Incidence rates, ranging from 28% to 56% within two years post-operation, exhibit variability, partly due to diverse presentations and potential underreporting by patients. The psychological impact of cardiac surgery often leads patients to normalize enduring pain, delaying the identification of chronic post-sternotomy pain.

The multifaceted etiology of CPSP after sternotomy remains incompletely understood. Factors such as neural sensitization during the acute phase, neuropathy from nerve entrapment or injury during surgery, musculoskeletal trauma from incisions, sternal complications, and infections contribute to this complex pain landscape. Inadequate management of acute perioperative pain can trigger central sensitization, a process-altering spinal pain pathway, and predispose individuals to hyperalgesia and chronic pain. Thus, effective acute pain control not only alleviates immediate postoperative discomfort but also potentially averts the onset of chronic pain.

Traditionally, opioids like fentanyl and morphine have been primary choices for post-cardiac surgery pain relief. However, their use is associated with dose-related side effects such as nausea, respiratory issues, chronic opioid dependence, and increased chronic pain risk. Implementing a multimodal approach, including NSAIDs, proves challenging due to bleeding and renal complications post-cardiac surgery. In contrast, regional analgesia offers an opioid-sparing alternative. Parasternal regional blocks like the pectointercostal fascial plane block (PIFB) present a low-risk option and have demonstrated efficacy in alleviating acute post-sternotomy pain.

Addressing this, a prospective, double-blinded randomized controlled trial aimed to evaluate whether a PIF block could provide effective perioperative analgesia and potentially mitigate the incidence of CPSP in patients undergoing sternotomy for cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA 3 risk score patients scheduled for elective open heart surgery

Exclusion Criteria:

* Emergent surgery
* Previous thoracotomy
* LVEF <30
* Patients with psychiatric disorders
* Presence of hematological disease
* Patients with alcohol-drug addiction
* Patients who use daily opioids for any reason
* Chronic analgesic use
* Allergy to local anesthetics
* BMI >40

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-01-18 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
chronic pain | 3 months
  Postoperative chronic pain will be evaluated using brief pain inventory at 3 months after cardiac surgery. Brief Pain Inventory is a questionnaire designed to capture both pain intensity and the amount of interference that pain has on functioning. Pain intensity is measured with four items (worst, least, on average, and currently). Interference is measured with seven items, including general activity, mood, walking, work (including paid and household work), relations with others, sleep, and enjoyment of life. The patient answers the items on a scale of 0-10, the highest number indicating the worst imaginable pain for intensity items and complete interference for interference items.

SECONDARY OUTCOMES:
Time to extubation | 24 hour
  After the operation, the time until the patient is extubated will be recorded.
Postoperative pain score | 72 hour
  Pain levels will be evaluated with the visual analog scale (VAS) at 0, 3, 6, 12, 24, 36, 48, and 72 hours after extubation. VAS use numbers to rate pain from 0 (no pain) to 10 (worst pain).
Postoperative nausea and vomiting (PONV) | 72 hour
  The patients will be verbally evaluated according to a descriptive five-point PONV scale at 0, 3, 6, 12, 24, 48 and 72 hours after extubation.
Length of stay in the ICU | 7 day
  The time from admission to the ICU to the time of discharge to the hospital ward; during the hospital stay, an average of 7 days.
The number of patients who required rescue analgesic | 72 hour
  The number of patients who require rescue analgesic will be recorded at 0, 3, 6, 12, 24, 36, 48, and 72 hours after extubation.

CONTACTS AND LOCATIONS:
Locations (1):
- Betul Kozanhan, Konya, Turkey (Türkiye)